CLINICAL TRIAL: NCT02952560
Title: A Comparative Study of Ultrasound Versus CT Measurement of Tongue and Oral Cavity Size: Validation of Sonographic Technique
Brief Title: A Comparative Study of Ultrasound Versus CT Measurement of Tongue and Oral Cavity Size
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0791-AE
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2016-10

CONDITIONS: Ultrasound Airway Imaging in Determining the Oral Cavity and Tongue Size
Keywords: Ultrasound; Computed Tomography; Oral cavity size; The Mallampati classification
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- High resolution CT Scan of the head and neck: Patients scheduled for high resolution computerized tomography (CT scan) of the head and neck as part of their medical investigation of thyroid or laryngeal disorders will be recruited for this study.
  Interventions: Other: Ultrasound scan

INTERVENTIONS:
Other: Ultrasound scan — Ultrasound scanning examinations will be performed twice (pre-CT scan and post CT-scan). Each examination will be performed by two observers who are blinded to each other's measured values.Patients will be asked to place a small sip of water (20 mL)in their mouth and keep the mouth open during the imaging. A second ultrasound examination of each patient by the two observers will be performed after the CT-scan.

SUMMARY:
Difficulty in managing the airway is the single most important cause of major anesthesia-related morbidity and mortality. The currently used clinical method of predicting airway difficulty used by anesthetists is limited and not very highly sensitive or specific. Any additional bedside method that increases its specificity and sensitivity would be valuable. This project is designed to study and measure the tongue thickness and oral cavity height by using an ultrasound scan and comparing them with the same measurements obtained by CT scan. These will also be compared to a more complicated measurements used in previous studies to investigate any correlation with the currently used clinical methods. This information will help us decide if ultrasound may help Anesthesiologists assess difficulties in airway management in a more accurate, precise and reliable simpler method.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 80 Years
* Gender: Both males and females are eligible for the study
* ASA I-III
* Scheduled for CT-scan of the head and neck as part of medical investigation (for test validation part)

Exclusion Criteria:

* Volunteer/ patient refusal
* Language Barrier
* Known oropharyngeal, laryngeal or head and neck disease or cancers
* Multiple amalgam fillings of the teeth
* Past history of oral or head and neck surgical procedures
* Past history of burns or radiotherapy of the head and neck region
* Presence of any scars, sinuses, infection, swelling, cysts in the head and neck region

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for high resolution computerized tomography (CT scan) of the head and neck as part of their medical investigation of thyroid or laryngeal disorders will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Validity of the assumption that ratio of "tongue thickness/oral cavity height" is a good estimate of the ratio "tongue volume/oral cavity volume" as measured by CT scan. | 2012-2013
Validity of ultrasound measurement of the two airway parameters (tongue thickness and height of oral cavity) against CT measurements of the same parameters. | 2012-2013

SECONDARY OUTCOMES:
Reproducibility of the ultrasound measurements | 2012-2013
Correlating ultrasound measured values with Mallampati scores | 2012-2013

CONTACTS AND LOCATIONS:
Overall Officials: Vincent W.S Chan, MD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Savva D. Prediction of difficult tracheal intubation. Br J Anaesth. 1994 Aug;73(2):149-53. doi: 10.1093/bja/73.2.149. PMID 7917726
- [Background] Werner SL, Smith CE, Goldstein JR, Jones RA, Cydulka RK. Pilot study to evaluate the accuracy of ultrasonography in confirming endotracheal tube placement. Ann Emerg Med. 2007 Jan;49(1):75-80. doi: 10.1016/j.annemergmed.2006.07.004. Epub 2006 Oct 2. PMID 17014927
- [Background] Lakhal K, Delplace X, Cottier JP, Tranquart F, Sauvagnac X, Mercier C, Fusciardi J, Laffon M. The feasibility of ultrasound to assess subglottic diameter. Anesth Analg. 2007 Mar;104(3):611-4. doi: 10.1213/01.ane.0000260136.53694.fe. PMID 17312218
- [Background] Tsui BC, Hui CM. Sublingual airway ultrasound imaging. Can J Anaesth. 2008 Nov;55(11):790-1. doi: 10.1007/BF03016357. No abstract available. PMID 19138924